CLINICAL TRIAL: NCT05500287
Title: Effect of Virtual Care Given To Child Patients With Asthma On Disease Management And Quality
Brief Title: Virtual Care In Pediatric Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Merve Gümüş, Researcher in the Nursing Faculty, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB.E.57802
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Asthma in Children
Keywords: Virtual Care
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Care Group (Experimental): Children in virtual care group (VCG) were given distance asthma education for the first month. The education was given in groups of 5-6 children. Also, short videos were taken by the researcher on how to use medications and nebulizers and were shown in Zoom meetings. The education and videos were prepared by scanning the current literature and expert opinion was obtained from 2 experts in nursing education, 2 experts in pediatric nursing and a expert in the pediatric allergy field. Children and families sent asthma diaries to the researcher every 4 weeks. At the end of the first, third and sixth months, data from asthma diaries were collected via Google Forms. The Pediatric Asthma Child Quality of Life Scale score was also collected through Google Forms at the beginning and end of the sixth month. The patients received support from the researcher on case management via telephone or video call 24/7. Case management was multidisciplinary (a nurse and a specialist).
  Interventions: Other: Virtual Care
- Control Group (No Intervention): Children and families who in the control group (CG), sent asthma diaries to the researcher every 4 weeks. At the end of the first, third and sixth months, data from asthma diaries were collected via Google Forms. The Pediatric Asthma Child Quality of Life Scale score was also collected through Google Forms at the beginning and end of the sixth month. In the CG, the education routinely given by the physician during the outpatient clinic visits continued in the same way. In the name of equality of opportunity, training presentations and videos were shared with the CG at the end of the study. Also, the training presentation was converted into a booklet (videos were added to the booklet in the form of QR codes) and delivered to the clinic in printed form.

INTERVENTIONS:
Other: Virtual Care — Children in the virtual care group had distance asthma education, case management and virtual care
  Arms: Virtual Care Group

SUMMARY:
The purpose of this study was to determine the impact of virtual care for children with asthma on the disease management and quality of life of children with asthma.

DETAILED DESCRIPTION:
After children were randomized by protocol number, they completed the child information form, the quality of life scale of the child with asthma, and the asthma control test at the first interview. PEF meter and asthma diary were given at the first interview. Children in the virtual care group received online training in four modules within the first month.The virtual group provided counseling services by phone and video conference for six months. The control group received the standard care provided in the clinic. Asthma diary data were collected from both groups at the end of each month

ELIGIBILITY:
Inclusion Criteria:

* having a smartphone or tablet with internet connection, parents and patient willing to maintain a daily log of symptoms and medication use

Exclusion Criteria:

* Children who had mental problems, had not attended at least one of the training and did not send at least one month of their asthma diary were excluded from the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in symptom number | first, third and the sixth month
  The children were given a asthma diary to track their daily symptom of asthma. Asthma diary includes symptoms of wheezing, cough, activity limitation, sleep disturbance and response fo the use of rescue medication. The diary includes also peakflow meter values for two times per day. A sympyom day means any day for which child recorded any symptom, or reported the use of rescue medication. Children and families kept an asthma diary throughout the study and sent it to the researcher every 4 weeks

SECONDARY OUTCOMES:
Change from baseline in quality of life | Baseline and sixth month
  The Pediatric Asthma Child Quality of Life Scale score was collected through internet

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We don't plan to make IPD available to other researchers.